CLINICAL TRIAL: NCT06632106
Title: In Which Tumor Burden Range Does Advanced Hepatocellular Carcinoma Patients Benefit More from Hepatic Arterial Infusion Chemotherapy Plus Immune Checkpoint Inhibitors and Tyrosine Kinase Inhibitors Than Immune Checkpoint Inhibitors Plus Tyrosine Kinase Inhibitors? a Multi-center, Retrospective, Propensity Score Matching Study
Brief Title: HAIC in Combination with Immune Checkpoint Inhibitors and Tyrosine Kinase Inhibitors for Advanced HCC
Status: Active, not recruiting | Type: Observational
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Haibo Shao, Professor, MD, PhD, First Hospital of China Medical University
Other Study IDs: NICER024
Record Dates: First submitted 2024-10-06; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Hepatic Arterial Infusion Chemotherapy; Tyrosine Kinase Inhibitor; Immune Checkpoint Inhibitors; Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Tyrosine Kinase Inhibitors; Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- HAIC plus TKIs and ICIs: Each patient should receive at least 2 cycles of HAIC and 1cycles of TKIs plus ICIs. The interval between HAIC and TKIs plus ICIs should be within 2 weeks.
  Interventions: Procedure: hepatic artery infusion chemotherapy; Drug: Tyrosine kinase inhibitor (TKIs); Drug: Immune Checkpoint Inhibitors
- TKIs plus ICIs: Each patient should receive at least 2 cycles of ICIs. The interval between TKIs and ICIs should be within 2 weeks.
  Interventions: Drug: Tyrosine kinase inhibitor (TKIs); Drug: Immune Checkpoint Inhibitors

INTERVENTIONS:
Procedure: hepatic artery infusion chemotherapy — Hepatic arterial infusion chemotherapy including FOLFOX and RALOX
  Groups: HAIC plus TKIs and ICIs
Drug: Tyrosine kinase inhibitor (TKIs) — TKIs including Lenvatinib, Sorafenib, Apatinib, Donafenib, Bevacizumab
Drug: Immune Checkpoint Inhibitors — ICIs including Camrelizumab, Sintilimab, Tislelizumab, Pembrolizumab, Atezolizumab

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of hepatic arterial infusion chemotherapy (HAIC) in combination with PD-1 inhibitors and Lenvatinib in patients with different tumor burden advanced-stage hepatocellular carcinoma (HCC) with portal vein tumor thrombus (PVTT).

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of HCC confirmed by radiology, histology, or cytology;
2. Barcelona Clinic Liver Cancer (BCLC) stage C with the presence of portal vein tumor thrombus;
3. Has not received any previous systemic therapy for HCC (including chemotherapy, molecularly targeted therapy, immunotherapy);
4. Both TKIs and ICIs patients received only include marketed drugs but are not limited to HCC approval;
5. HAIC was performed after the first TKIs/ ICIs treatment or before treatment;
6. Received at least 2 cycles of HAIC or ICIs treatments；
7. Has repeated measurable intrahepatic lesions;
8. Child-Pugh class A or B.

Exclusion Criteria:

1. Patients who took systemic anti-tumor treatments before the combination therapy;
2. With other malignant tumors;
3. Unable to meet criteria of combination timeframe described above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced HCC with PVTT who received HAIC in combination with TKIs and ICIs under real-world practice conditions.
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to approximately 2 years
  The OS is defined as the time from the initiation of any combination treatment to death due to any cause.

SECONDARY OUTCOMES:
Progression free survival(PFS) | Up to approximately 2 years
  The PFS is defined as the time from the initiation of any combination treatment to the first documented progressive disease (according to RECIST1.1) or death due to any cause, whichever occurs first.
Objective response rate(ORR) per RESCIST 1.1 | Up to approximately 2 years
  The ORR is defined as the proportion of patients with a documented complete response(CR) or partial response(PR) per RECIST 1.1.
ORR of PVTT | Up to approximately 2 years
  The ORR is defined as the proportion of patients with a documented CR or PR of PVTT.
Adverse event(AE) per Common Terminology Criteria for Adverse Events(CTCAE) 5.0 | Up to approximately 2 years
  The percentage and degree of patients who experience at least one AE, whether or not considered related to the treatment, according to CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of China medical university, Shenyang, Liaoning, China